CLINICAL TRIAL: NCT06081660
Title: Advance Care Planning for Older Latinos With Chronic Illness: A Feasibility Study
Brief Title: Advance Care Planning for Older Latinos With Chronic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Frances Nedjat-Haiem, Associate Professor, San Diego State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-2020-0175
Record Dates: First submitted 2022-11-21; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Patient Engagement; End of Life; Chronic Disease; Communication
Keywords: Latino; Advance Care Planning; Advance Directive
MeSH Terms: conditions — Patient Participation; Death; Chronic Disease; Communication

STUDY DESIGN:
Intervention Model Description: 2 x 2 mixed factorial design, pre-test/posttest variables to examine impact on ACP
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACP education (Active Comparator): ACP education consisting of
  * a brief social work screening,
  * an educational pamphlet,
  * advance directive forms (in English and Spanish), and
  * community resource materials (i.e., handout)
  Interventions: Behavioral: ACP-I Plan
- ACP education plus counseling (Experimental): ACP education plus counseling consisting of
  * a brief social work screening,
  * an educational pamphlet,
  * advance directive forms (in English and Spanish), and
  * community resource materials (i.e., handout);
  * motivational interviewing
  * decisional support, and
  * patient navigation to address barriers
  Interventions: Behavioral: ACP-I Plan

INTERVENTIONS:
Behavioral: ACP-I Plan — ACP-I Plan consisting of education, counseling, decisional support, and patient navigation

SUMMARY:
The goal of this study is to test the feasibility of a randomized controlled trial to learn about implementation of an intervention model, Advance Care Planning I Plan (ACP-I Plan), among older Latinos with chronic illnesses in community settings.

DETAILED DESCRIPTION:
The goal of this study is to test the feasibility of a randomized controlled trial to learn about implementation of an intervention model, Advance Care Planning I Plan (ACP-I Plan), among older Latinos with chronic illnesses in community settings.

The questions of this study seek to explore implementation of the intervention model:

1. To evaluate feasibility, acceptability, and preliminary impact of ACP-I Plan to improve AD documentation and increase engagement in ACP communication with family and providers among older Latinos with chronic diseases (cancers and non-cancers); and
2. To evaluate implementation of ACP-I Plan in a community setting and examine further need for adaption.

Participants will be randomized into two groups:

1. ACP education consisting of

   * a brief social work screening,
   * an educational pamphlet,
   * advance directive forms (in English and Spanish), and
   * community resource materials (i.e., handout); and
2. ACP education plus counseling consisting of

   * motivational interviewing
   * decisional support, and
   * patient navigation to address barriers We anticipate that ACP-I Plan will be feasibly and acceptable. Participants who receive ACP-I Plan will show 1) greater likelihood of documenting an AD, 2) greater importance of and concern for engaging in ACP communication with family members and providers, and 3) reduced distress at 4-week post intervention.

ELIGIBILITY:
Inclusion Criteria:

* 50 years old or older
* Latino/Latina or Hispanic?
* Have 1 or more chronic health conditions

Exclusion Criteria:

* Schizophrenia
* Schizoaffective Disorder
* Dementia
* Alzheimer's disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-04-16 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility | 12 months
  Feasibility
  We use benchmarks for feasibility.
  1. Number of Participants Recruited, and screening no more than 100 participants,
  2. tracking numbers of participants consented into the study,
  3. percent refused to participate and dropout, amount of time to screen participants and complete a baseline survey once consented into the study,
  4. ACP-I Plan intervention delivered for the first session <2 weeks from their recruitment and randomization date and second session <4 weeks from recruitment,
  5. identify missing data.
  6. Track the number of participants who indicate they returned a completed AD to their provider and/or talked with a family member regarding ACP.
Satisfaction with intervention | 1 month
  Acceptability of the intervention
  Satisfaction survey questions includes 14 questions using "I" statements and a 5-point Likert scale: Strongly Disagree to Strongly Agree). Improved scores at follow up indicate satisfaction of information delivery.
  Reference
  Lyon ME, Garvie PA, Briggs L, He J, McCarter R, D'Angelo LJJJopm. Development, feasibility, and acceptability of the Family/Adolescent-Centered (FACE) Advance Care Planning intervention for adolescents with HIV. 2009;12(4):363-372.
Retention and Attrition Rates | 12 months
  Feasibility of recruitment and retention

SECONDARY OUTCOMES:
Completion Rates | 1 month
  Self report yes/no completed an advance directive document.
  We use the method that Douglas & Brown (2002) used ask about completion of advance directives at 2 points, baseline and 1-month follow-up. Questions have yes/no [Y/N], responses.
  Reference Douglas R, Brown HN. Patients' attitudes toward advance directives. Journal of Nursing Scholarship.
  2002;34(1):61-65.
  We also use the Advance Directive Attitude Survey (ADAS) by Nolan has 16 items and asks questions (uses a 4-point Likert scale, Strongly Agree to Strongly Disagree with AD decision making). Sixteen questions are subscales and ask about: (a) opportunity for treatment choices, (b) effect of advance directives on the family, (c) effect of an AD on treatment, and (d) perception of illness.
  Nolan MT, Bruder M. Patients' attitudes toward advance directives and end-of-life treatment decisions. Nursing outlook. 1997;45(5):204-208.
Communication Readiness Provider | 1 month
  Barriers to ACP communication and readiness to talk with provider.
  We use a barrier scale developed to identify Barriers to Communication about Advance Care Planning (Nedjat-Haiem, 2022) which has 19 questions and uses a scale from 0 to 4, asking how much of a concern is this for you? Readiness to engage in communication about ACP will be assessed by three yes/no questions that ask about: (1) fear of death and dying, (2) difficulty engaging in EOL care communication, and (3) worry about illness severity.
  We also use a readiness scale (1-10) which asks: how ready are you to engage in ACP communication with your physician.
Communication Readiness Family | 1 month
  Self Report yes/no - Readiness to talk with a family member
  We also use one question to ask about about readiness using a scale (1-10) which asks: how ready are you to engage in ACP communication with your family member?

CONTACTS AND LOCATIONS:
Overall Officials: Ayala, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States